CLINICAL TRIAL: NCT03750071
Title: An Open-label, Phase I/II Multicenter Clinical Trial of VXM01 in Combination With Avelumab in Patients With Progressive Glioblastoma Following Standard Treatment, With or Without Second Surgery
Brief Title: VXM01 Plus Avelumab Combination Study in Progressive Glioblastoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vaximm GmbH (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VXM01-AVE-04-INT
Record Dates: First submitted 2018-10-26; First posted 2018-11-21 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VXM01/Avelumab (Experimental): Combination of VXM01, Ty21a transformed with a eukaryotic expression cassette encoding VEGFR-2, and anti-PD-L1 Checkpoint Inhibitor Avelumab
  Interventions: Biological: VXM01; Biological: Avelumab

INTERVENTIONS:
Biological: VXM01 — Ty21a transformed with a eukaryotic VEGFR-2 Expression Plasmid
  Other Names: Investigational VEGFR-2 DNA Vaccine
Biological: Avelumab — Monoclonal anti-PD-L1 Antibody
  Other Names: Bavencio

SUMMARY:
VXM01 in combination with avelumab in n=30 patients with progressive glioblastoma following standard treatment, with or without second surgery

DETAILED DESCRIPTION:
The trial is conducted as a multicenter, open-label, Phase I/II trial to evaluate the efficacy and safety of VXM01 in combination with avelumab in subjects with resectable and non-resectable progressive glioblastoma following tumor resection and radiochemotherapy containing temozolomide.

The trial will be performed in 30 subjects with progressive glioblastoma:

* 24 subjects who will not be candidates for a tumor re-operation (non-resectable subjects)
* 6 subjects who will be candidates for a tumor re-operation (resectable subjects) The trial, for each subject, will consist of a screening period, a treatment and observatioon phase of 60 weeks including, a treatment phase of up to 48 weeks with prime and boosting administrations of VXM01 in combination with avelumab and an observation phase of 12 weeks and with an end of trial visit at Week 60.

Subjects will receive VXM01 in combination with avelumab up to Week 48. The end of study (EoS) visit assessments will be performed Week 60.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able to understand and follow instructions during the trial
2. Ability and willingness to give written informed consent, signed and dated
3. Male or female subjects. Female subjects must be post-menopausal for at least 2 years or surgically sterile
4. Age ≥18 years
5. Histologically diagnosed intracranial supratentorial malignant glioma (glioblastoma WHO Grade IV)
6. Evidence of tumor progression by RANO criteria following at least one prior therapy regimen that must have contained radiation and chemotherapy with temozolomide, as measured by MRI

   - Radiotherapy must have been completed at least 3 months prior to the inclusion visit
7. Candidates for a tumor reoperation (for the resectable arm [n=6] only)

   - Neurosurgical intervention should be postponable for 30 days
8. Adequate bone marrow function including: Absolute neutrophil count (ANC) ≥1,500/mm3 or ≥1.5 x 109/L; Platelets ≥ 100,000/mm3 or ≥100 x 109/L; Hemoglobin ≥ 9 g/dL (may have been transfused); INR <1.5x ULN. Subjects with documented benign cyclical neutropenia are allowed if WBC count is ≥ 1.5 × 109/L with absolute neutrophil count ≥ 1.0 × 109/L and appropriate hematology parameters: leukocytes ≥4.0 x 109 / L, lymphocytes ≥0.6 x 109/L
9. Adequate hepatic function defined by a total bilirubin level ≤ 1.5 × the upper limit of normal range (ULN), an aspartate aminotransferase (AST), level ≤ 2.5 × ULN, and an alanine aminotransferase (ALT) level ≤ 2.5 × ULN or, for subjects with documented metastatic disease to the liver, AST and ALT levels ≤ 5 × ULN. Subjects with documented Gilbert disease are allowed if total bilirubin ≤ 3 x ULN
10. Adequate renal function defined by an estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula
11. Patients must be able to undergo MRI
12. Absence of active bacterial infection requiring antibiotic treatment
13. Karnofsky performance status ≥70
14. Primary tumor samples available for pathology review, central detection of T-cell responses in the peripheral blood and in the tumor tissue
15. No medical or social conditions that may interfere with trial outcome and follow-up

Exclusion Criteria:

1. Cardiovascular disease defined as:

   1. Uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg)
   2. Arterial thromboembolic event within 6 months before trial entry, including:

   i. Myocardial infarction ii. Unstable angina pectoris iii. Cerebrovascular accident iv. Transient ischemic attack
2. Congestive heart failure New York Heart Association grade III to IV
3. Serious ventricular arrhythmia requiring medication and arrhythmias requiring Implantable Cardioverter Defibrillator (ICDs)
4. Clinically significant peripheral artery disease > grade 2b according to Fontaine
5. History of intracranial hemorrhage
6. Hemoptysis within 6 months before trial entry
7. Known oesophageal varices
8. Upper or lower gastrointestinal bleeding within 6 months before inclusion (Day 0)
9. Significant traumatic injury or surgery within 4 weeks before trial entry
10. Non-healing wound, incomplete wound healing, bone fracture or gastrointestinal ulcers within three years before inclusion, or positive gastroscopy within 3 months before inclusion
11. Gastrointestinal fistula
12. Thrombolysis therapy within 4 weeks before trial entry
13. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that based on the investigator's judgement provides a reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the trial results or render the patient at high risk for treatment complications
14. Previous malignant disease (other than the tumor disease for this trial) within the last 5 years (except adequately treated non-melanoma skin cancers, carcinoma in situ of skin, bladder, cervix, colon/rectum, breast, or prostate) unless a complete remission without further recurrence was achieved at least 2 years prior to trial entry and the subject was deemed to have been cured with no additional therapy required or anticipated to be required
15. Prior organ transplantation, including allogeneic stem cell transplantation
16. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:

    1. Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
    2. Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) are acceptable
17. History of uncontrolled intercurrent illness including but not limited to uncontrolled diabetes (e.g., hemoglobin A1c ≥ 8%)
18. Known prior hypersensitivity to investigational product or any component in its formulations or any other drug scheduled or likely to be given during the trial, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5.0 Grade ≥ 3)
19. Persisting toxicity related to prior therapy (NCI CTCAE v5.0 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 AEs not constituting a safety risk based on investigator's judgment are acceptable
20. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormalities that may increase the Risk associated with trial participation or trial treatment administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into this trial
21. Active infection requiring systemic therapy
22. Known history of human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome or multi-drug resistant gram-negative bacteria
23. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
24. Women of childbearing potential
25. History of serious ophthalmological diseases, e.g. optic neuropathy, retinal detachment, uveitis Prior and concomitant medication
26. Treatment in any other clinical trial within 30 days or within 5 half lives of any prior treatment, before screening
27. Any other condition or treatment that, in the opinion of the investigator, might interfere with the trial or current drug or substance abuse
28. Chronic concurrent therapy within 2 weeks before and during the treatment period with:

    1. Corticosteroids (except steroids up to equivalent of dexamethasone 4 mg daily dose)
    2. Immunosuppressive agents
    3. Antibiotics
    4. Bevacizumab or any other anti-angiogenic treatment
    5. Any other anti-cancer therapy or concurrent anticancer treatment, for example, cytoreductive therapy, radiotherapy [with the exception of palliative short course, limited field (ie, ≤ 10 fractions and ≤ 30% bone marrow involvement or per institutional standard) radiotherapy, which may be administered during the study. However dosing must be suspended at least 14 days prior to the start of radiotherapy and must not be resumed until at least 14 days after the last radiotherapy fraction], immune therapy, or cytokine therapy, except for erythropoietin
    6. Administration of live vaccines (other than VXM01) within 30 days prior to study treatment Other
29. Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines (other than VXM01)
30. Inability to understand the protocol requirements, instructions and trial-related restrictions, the nature, scope, and possible consequences of the trial
31. Unlikely to comply with the protocol requirements, instructions and trial-related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits, and improbability of completing the trial
32. Legal incapacity or limited legal capacity
33. Any condition which results in an undue risk for the patient during the trial participation according to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-emerging adverse events (safety and tolerability of VXM01 in combination with avelumab) | Up to 60 weeks after first IMP administration
  AEs listed together with information on onset, duration, severity, seriousness, relationship to the study drug, relationship to chemotherapy and to the underlying disease, outcome, and action taken. Frequency tables by System Organ Class and preferred term.

SECONDARY OUTCOMES:
Clinical response as assessed by time to progression (TTP) | Up to 60 weeks after first IMP administration
  TTP is defined from the day of trial entry to the day of local tumor progression based on MRI (in days)
Clinical response as assessed by progression free survival (PFS) | Up to 60 weeks after first IMP administration
  PFS is defined from the day of trial entry to the day of local tumor progression or recurrence after reoperation, based on MRI, or further positive biopsy, or the day of death of any cause. Subjects free of progression/recurrence will be censored at the day of last tumor assessment (in days)
Clinical response as assessed by recurrence-free survival after re-operation (RFS) | Up to 60 weeks after first IMP administration
  RFS is defined from the day of trial entry to the day of recurrence after reoperation, based on MRI (in days)
Clinical response as assessed by Overall Survival (OS) | Up to 60 weeks after first IMP administration
  OSOS will be defined by death of any cause and subjects alive at trial end will be censored at last contact day (in days)
Best overall response (OR) on MRI according to iRANO in subjects with or without surgery prior to trial entry (up to re-operation) | Up to 60 weeks after first IMP administration
  The proportion of subjects with OR will be estimated together with 95% confidence intervals constructed using the binomial Distribution (in %)
Duration of Response (DoR) on MRI according to iRANO in subjects with or without surgery prior to trial entry (up to re-operation) | Up to 60 weeks after first IMP administration
  The DoR on MRI according to iRANO will be summarized descriptively for the two subgroups and illustrated using a Kaplan-Meier plot

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Wick, MD, Principal Investigator — University Clinics Heidelberg
Locations (2):
- Germany (2):
  - Neurology Clinic and National Center for Tumor Diseases, Heidelberg
  - Neurology Clinic, Mannheim

IPD SHARING:
Plan to Share IPD: No